CLINICAL TRIAL: NCT07401212
Title: The Impact of Chronic Consumption of Prebiotics on Cognitive and Affective Outcomes, Gut Microbiome Diversity and Composition in 3-5 Year Olds: a Double-blind Placebo-controlled, Parallel-groups Randomised Controlled Trial
Brief Title: GUTLINK4KIDS Intervention
Acronym: GUTLINK4KIDS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Beneo GmbH (Industry)
Responsible Party: Principal Investigator, Piril Hepsomali, Principle Investigator, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UREC25_38
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Temperament; Sleep; Cognition; Emotion Regulation
Keywords: prebiotics; emotion regulation; gut microbiome diversity; children; relative abundance; sleep; internalising symptoms; externalising symptoms
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prebiotic (powder) (Experimental): Children will consume two (one in the morning and one in the evening) 2.5g of prebiotic sachets a day (mixed with food and drink).
  Interventions: Dietary Supplement: Prebiotic powder
- Matched placebo (powder) (Placebo Comparator): Children will consume two (one in the morning and one in the evening) 2.5g of placebo sachets a day (mixed with food and drink).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Prebiotic powder — 5g of prebiotic fibre
  Arms: Prebiotic (powder)
Dietary Supplement: Placebo — 5g of placebo
  Arms: Matched placebo (powder)

SUMMARY:
This study aims to investigate the chronic effects of prebiotic consumption on cognitive, behavioural and gut microbiome outcomes in children aged 3-5 years.

DETAILED DESCRIPTION:
This study will employ a double-blind, randomised, placebo-controlled parallel design to investigate the chronic effects of 8-week-long prebiotic consumption on cognitive, behavioural, and gut microbiome, outcomes in 3-5-year-old children with insufficient fibre intake (less than the average 10.4g/day in 18-47-month-olds and less than 12.6g/day in 48-60-month-olds). One hundred and six participants will be randomised to Intervention or Placebo groups where they will be consuming 5g of prebiotic fibre or 5g of placebo (matched placebo powder) per day for 8-weeks. Outcome measures will be acquired before and after a 8-week chronic supplementation. These will include cognitive and behavioural outcomes of the parents and children. In addition, stool samples will be collected at the baseline and at week 8 to assess microbiome diversity and composition. Additionally, after 4-weeks of wash-out, at 12 weeks, parents will be asked to completed online questionnaires assessing cognitive and behavioural outcome of their children.

ELIGIBILITY:
Inclusion Criteria:

* Parents (18 years and over) of generally healthy children aged 3-5-years-old (36-71 months) with lower dietary fibre intake than the recommended daily amount (10.4g/day in 18-47-month-olds and less than 12.6g/day in 48-60-month-olds).

Exclusion Criteria:

* Children with a significant acute or chronic co-existing illness (including inflammatory bowel disease, functional gastrointestinal disorders, coeliac disease etc, neurodevelopmental, immunological, psychiatric, or metabolic disorders.
* Children who have taken any pre/probiotic supplements or antibiotic treatment within the 4 weeks prior to enrolment.
* Children with food allergies and intolerances

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 106 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Child Behaviour Checklist Ages 1.5-5 | This measure will be taken at baseline (pre intervention), week 8 (post intervention) and week 12 (after 4-week wash-out)
  Parents will be asked to complete this validated measure that includes 100 items that assesses a child's emotional, behavioral, and social problems.

SECONDARY OUTCOMES:
Emotion Regulation Skills Questionnaire | This measure will be taken at baseline (pre intervention), week 8 (post intervention) and week 12 (after 4-week wash-out)
  Parents will be asked to complete this measure that includes 52 items that assesses a child's adaptive and maladaptive emotion regulation skills.
Childhood Autism Spectrum Test | This measure will be taken at baseline (pre intervention), week 8 (post intervention) and week 12 (after 4-week wash-out)
  Parents will be asked to complete this measure that includes 44 items that assesses a child's developmental differences in social and communication functioning
Bristol Stool Chart | This measure will be taken at baseline (pre intervention), week 8 (post intervention) and week 12 (after 4-week wash-out)
  Parents will be asked to complete this measure that includes 1 item that assesses a child's stool consistency.
Gut microbiome diversity | This measure will be taken at baseline (pre intervention) and week 8 (post intervention).
  Children's stool samples will be collected to measure gut microbiome diversity. Indices of alpha and beta diversity will be analysed (16s sequencing).
Gut microbiome composition | This measure will be taken at baseline (pre intervention) and week 8 (post intervention).
  Children's stool samples will be collected to measure gut microbiome composition (genus and species) (16s sequencing).

OTHER OUTCOMES:
Attentional Control Scale | This measure will be taken at baseline (pre intervention) and week 8 (post intervention).
  Parents will be asked to complete this measure that includes 20 items that assesses their own attentional control.
Difficulties in Emotional Regulation Scale | This measure will be taken at baseline (pre intervention) and week 8 (post intervention).
  Parents will be asked to complete this measure that includes 36 items that assesses their own emotion regulation skills.
Patient Health Questionnaire-8 | This measure will be taken at baseline (pre intervention) and week 8 (post intervention).
  Parents will be asked to complete this measure that includes 8 items that assesses their own depressed mood.
Generalised Anxiety Disorder-7 | This measure will be taken at baseline (pre intervention) and week 8 (post intervention).
  Parents will be asked to complete this measure that includes 7 items that assesses their own anxious mood.
Child-Parent Relationship Scale | This measure will be taken at baseline (pre intervention) and week 8 (post intervention).
  Parents will be asked to complete this measure that includes 30 items that assesses their relationship with their child/children.
Scottish Collaborative Group Child VC2 Food Frequency Questionnaire | This measure will be taken at baseline (pre intervention).
  Parents will be asked to complete this measure that assesses their child's habitual food intake.
Child Eating Behaviour Questionnaire | This measure will be taken at baseline (pre intervention).
  Parents will be asked to complete this measure that assesses their child's eating behaviour.
Dietary recall | This measure will be taken during screening and at week 8 (post intervention).
  This measure will be used to screen participants. Parents will be asked to complete this measure that assesses their child's food intake. Children with insufficient fibre intake (less than the average 10.4g/day in 18-47-month-olds and less than 12.6g/day in 48-60-month-olds) will be eligible for the study.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, School of Psychology and Clinical Languages, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No